CLINICAL TRIAL: NCT03841474
Title: The Changes in Functional Recovery and Brain Neurotrophic Factor Six Months After Percutaneous Coronary Intervention in Cardiovascular Patients With Depression
Brief Title: The Recovery of Cardiovascular Patients With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Responsible Party: Principal Investigator, Sara Medved, Principal Investigator, Klinički Bolnički Centar Zagreb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBC Zagreb CoroDep
Record Dates: First submitted 2019-01-13; First posted 2019-02-15 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease; Depression; Cardiovascular Diseases
Keywords: Brain derived neurotrophic factor; BDNF; Psychosocial indicators; Depression; Cardiovascular disease
MeSH Terms: conditions — Coronary Artery Disease; Depression; Cardiovascular Diseases | interventions — Sertraline; Escitalopram; Methods

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to intervention group if they have symptoms of depression, i.e. to control group if they do not show depressive symptoms.
  A psychiatrist will then, according to clinical impression, prescribe either sertraline or escitalopram to intervention group (i.e. groups). Both groups (sertraline and escitalopram) will be described as one intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention I (Experimental): Psychiatric treatment with sertraline (range from 50 mg/day to 200mg/day according to clinical appearance) of cardiovascular patients after PCI with mild, moderate or severe depression
  Interventions: Drug: Psychiatric treatment with sertraline
- Control (No Intervention): Cardiovascular patients after PCI without depressive symptoms and without the need for psychiatric intervention
- Intervention II (Experimental): Psychiatric treatment with escitalopram (range from 10 mg/day to 20 mg/day according to clinical appearance) of cardiovascular patients after PCI with mild, moderate or severe depression
  Interventions: Drug: Psychiatric treatment with escitalopram

INTERVENTIONS:
Drug: Psychiatric treatment with sertraline — Psychiatric treatment with sertraline (range from 50 mg/day to 200mg/day according to clinical appearance) of newly recognized depression in patients after PCI
  Other Names: Intervention I
  Arms: Intervention I
Drug: Psychiatric treatment with escitalopram — Psychiatric treatment with escitalopram (range from 10 mg/day to 20 mg/day according to clinical appearance) of newly recognized depression in patients after PCI
  Other Names: Intervention II
  Arms: Intervention II

SUMMARY:
Cardiovascular disease increases the risk of depression and vice versa. Many cardiovascular patients are subjected to percutaneous coronary intervention (PCI). Potential biomarkers for the development, the course and the recovery of both diseases are in the focus of interest of many studies. One of the biomarkers that stands out is brain derived neurotrophic factor (BDFN). BDNF plays a significant role in regulating vascular growth and repair but also stimulates the survival, differentiation, and conservation of neurons.

The aim of the study is to detect the depression in patients undergoing PCI and to determine the impact of psychiatric treatment on the functional recovery and on the changes of BDNF.

DETAILED DESCRIPTION:
It has been shown that cardiovascular disease increases the risk of depression and vice versa. A significant proportion of cardiovascular diseases are coronary artery disease; most of these patients are subjected to percutaneous coronary intervention (PCI). That population of patients, which is under greater risk of depression, has been passing through the health system without adequate management of psychiatric difficulties. Despite the abundance of the data regarding the concomitancy of cardiovascular disease and depression, potential biomarkers for the development, the course and the recovery of both diseases are still in the focus of interest of many studies. One of the biomarkers that stands out is brain derived neurotrophic factor (BDFN). BDNF plays a significant role in regulating vascular growth and repair but also stimulates the survival, differentiation, and conservation of neurons. Its' serum level is reduced in cardiac failure and acute coronary syndrome, and indicates a higher risk of coronary incident in angina pectoris. BDNF is also reduced in depression, but increases during a pharmacological treatment along with the clinical improvement.

Therefore the aim of the study is to detect the occurrence of depression in patients undergoing PCI and to determine the impact of psychiatric treatment on the functional recovery of those patient and the correlation with the changes of serum levels of BDNF.

This represents the objectivization of the tertiary type of prevention intervention for recovery of cardiovascular patients who are currently passing through the investigator's health system with unrecognized psychiatric comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* patients on day of percutaneous coronary intervention due to angina pectoris or myocardial infarction
* without antidepressant drugs or major tranquilizers more than one year

Exclusion Criteria:

* symptoms of myocardial infarction lasting more than 12 hours
* left ventricle ejection function (LVEF) less than 40%
* earlier presence of cardiomyopathy
* acute infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Montgomery Asberg Depression Scale (MADRS) at 6 months | baseline, six months
  A 10-item clinician-administered questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Ten questions rate the severity of symptoms on scale of 0 (not present), 2 (mild), 4 (moderate), and 6 (severe).
Change from Baseline Hamilton Rating Scale for Depression (HAM-D) at 6 months | baseline, six months
  Semi-structured interview with 17 questions, designed to measure the severity of depressive symptoms in patients with a primary depressive illness. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. A score of 0-7 is considered to be normal while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Change from Baseline Beck Depression Inventory (BDI) at 6 months | baseline, six months
  A 21-question multiple-choice self-report inventory, with each question having a set of four and more possible responses, ranging in intensity. A value of 0 to 3 is assigned for each answer and the total score represents the sum of the values. Higher total score indicates more severe depressive symptoms.

SECONDARY OUTCOMES:
Change from Baseline EuroQol Group 3-level version instrument (EQ-5D-3L) at 6 months | baseline, six month
  EQ-5D is a standardized instrument for measuring generic health status. Questionnaire has five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and all dimensions are described by 3 problem levels corresponding to patient response choices. In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale.
Change from Baseline The Global Registry of Acute Coronary Events (GRACE ACS Risk Model) at 6 months | baseline, six months
  Changes in GRACE ACS Risk Model of cardiovascular patients six months after PCI
Change from Baseline Duke Activity Status Index (DASI) at 6 months | baseline, six months
  The Duke Activity Status Index (DASI) is an a 12-item questionnaire assessment tool used to evaluate the functional capacity of patients with cardiovascular disease. Each item has a specific weight based on the metabolic cost. The final score ranges between zero and 58.2 points. The higher the score indicates better functional capacity.
Change from Baseline The Seattle Angina Questionnaire (SAQ-7) at 6 months | baseline, six months
  SAQ is a 19-item instrument that measures patient-reported symptoms, function and quality of life for patients with coronary artery disease. The answers patients give to the SAQ's questions are used to calculate scores in five scales: anginal stability, anginal frequency, physical limitation, treatment satisfaction and quality of life. Each scale is transformed to a score of 0 to 100, where higher scores indicate better functioning.
Changes of blood serum concentrations of brain derived neurotrophic factor (BDNF) at 6 months | baseline, six months
  Changes in the serum levels of BDNF six months after PCI in cardiovascular patients without and cardiovascular patients with depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Alma Mihaljević Peleš, Prof., Study Chair — Head of Department of Psychiatry
Locations (1):
- KBC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No